CLINICAL TRIAL: NCT03551977
Title: Cultural Adaptation and Evaluation of the "iCanCope With Pain" App Among Norwegian Adolescents Living With Pain
Brief Title: The Norwegian "iCanCope With Pain" App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Agder (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Erik Grasaas, Principal Investigator, University of Agder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1310 63221
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: A single-centre, RCT study design with two arms, one control group (N=56) and one intervention group (N=56).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive the iCanCope with Pain app with all five components: (I) symptom trackers for pain, sleep, mood, physical, and social function; (II) goal setting to improve pain and function; (III) coping toolbox of pain self-management strategies; (IV) social support; (V) age-appropriate pain education
  Interventions: Behavioral: iCanCope with Pain
- Control group (Active Comparator): The control group will receive the iCanCope with Pain control app with only the first self-registration component (I) symptom trackers for pain, sleep, mood, physical, and social function.
  Interventions: Behavioral: iCanCope with Pain control

INTERVENTIONS:
Behavioral: iCanCope with Pain — The participants are free to use the Norwegian iCanCope with Pain app as much as they want during the 8 week intervention period. The only support available is technical support.
  Arms: Intervention group
Behavioral: iCanCope with Pain control — The participants are free to use the Norwegian iCanCope with Pain control app as much as they want during the 8 week intervention period. The only support available is technical support.
  Arms: Control group

SUMMARY:
Background: Research evidence shows that prevalence of pain in adolescents is increasing and is therefore recognized as a growing health problem. Psychological interventions delivered remotely through the internet may reduce intensity or severity of pain among children and adolescents with chronic pain. The iCanCope with Pain program is an existing web- and mobile-based self-management program, which is developed as a multi-center study funded by the Canadian Institutes of Health Research and is based on identified health care needs and current best practices for pain self-management.

Objectives: The primary objectives are to describe the translation and cultural adaptation of the Norwegian version of the iCanCope with Pain mobile application and evaluate the effect in an upcoming randomized controlled trail with adolescents with chronic pain.

Study sample: 16-19-year-old adolescents with self-declared persistent and/or chronic pain. Recruited from high schools in Southern Norway.

Theoretical framework: Cognitive behavioral therapy (CBT) is explained by an integration of behavioral and cognitive theories of human behavior and psychopathology and is often the preferred treatment of choice for adolescents with different health disorders. The theoretical framework of CBT is integrated in the iCanCope with Pain app in terms of five components. The intervention group will receive the app with all five components: (I) symptom trackers for pain, sleep, mood, physical, and social function; (II) goal setting to improve pain and function; (III) coping toolbox of pain self-management strategies; (IV) social support; (V) age-appropriate pain education. The control group will receive the app with only the first self-registration component (I) symptom trackers for pain, sleep, mood, physical, and social function.

Methods: Both qualitative and quantitative data will be gathered for evaluating the Norwegian version of the iCanCope with Pain app. Usability testing are assessed in both laboratory settings and in field using observation, interviews and questionnaires, which provide necessary information for an upcoming randomized controlled trail (RCT). Outcomes will in the RCT be measured at baseline (mid-April) and after an 8 weeks intervention (mid-June).

The study is part of a PhD project.

ELIGIBILITY:
Inclusion Criteria:

1. 16-19-year-old adolescents
2. with persistent and/or chronic pain, weekly suffered and lasting 3 months or more based on subjective reporting
3. be able to read and understand Norwegian
4. have their own smartphone.

Exclusion Criteria:

1. Adolescents with cognitive disability or diseases, because of the risk of not correctly understanding the iCanCope with Pain program via self-report, goal setting and/or library reading.
2. Adolescents that have participated in the usability testing of the Norwegian iCanCope with Pain app
3. Adolescents with diagnoses from a pathological or medical origin (e.g hematology/oncology patients) will also be excluded because the program was not specifically designed for these pain groups.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Attrition rate | Baseline and 8-weeks
  Change in participants completed the post-questionnaire divided by the number of participants at baseline.
App engagement | Baseline to 8 weeks.
  Completion of daily symptom check-ins was used as a proxy for app engagement.

SECONDARY OUTCOMES:
Physical activity | Baseline and 8 weeks (post-intervention)
  Change in total score of the International Physical Activity Questionnaire (IPAQ). Higher values at post-intervention represent a better outcome.
Coping | Baseline and 8 weeks (post-intervention)
  Change in total score of the General Self-Efficacy Questionnaire Short Version (GSEQ). Higher values at post-intervention represent a better outcome.
Social participation | Baseline and 8 weeks (post-intervention)
  Change in total score of school absence (General Information Questionnaire). Lower values at post-intervention represent a better outcome.
Over-The-Counter (OTC) analgesics | Baseline and 8 weeks (post-intervention)
  Change in total score of OTC analgesics consumption (General Information Questionnaire). Lower values at post-intervention represent a better outcome.
Perceived social support from friends | Baseline and 8 weeks (post-intervention)
  Change in total score of the Perceived Social Support from friends Questionnaire (PSS). Higher values at post-intervention represent a better outcome.
Pain self-efficacy questionnaire | Baseline and 8 weeks (post-intervention)
  Change in total score of the Pain Self-Efficacy Questionnaire (PSEQ). Higher values at post-intervention represent a better outcome.
Anxiety and depression | Baseline and 8 weeks (post-intervention)
  Change in total score of the Hospital Anxiety and Depression Scale Questionnaire (HADS). Lower values at post-intervention represent a better outcome.
Global impression of change | After 8 weeks (post-intervention)
  Change in Patients' Global Impression of Change Scale (PGIC) from 1-7. Higher values at post-intervention represent a better outcome.
Health-related quality of life (HRQOL) | Baseline and 8 weeks (post-intervention)
  Change in total score of the Kidscreen 52 Questionnaire. Higher values at post-intervention represent a better outcome.
Pain experience | Baseline and 8 weeks (post-intervention)
  Change in total score of the Lubeck Pain Questionnaire (LPQ). Lower values at post-intervention represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Haraldstad, PhD, Principal Investigator — UiA
Locations (1):
- Erik Grasaas, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grasaas E, Helseth S, Fegran L, Stinson J, Smastuen M, Lalloo C, Haraldstad K. App-based intervention among adolescents with persistent pain: a pilot feasibility randomized controlled trial. Pilot Feasibility Stud. 2022 Jul 27;8(1):158. doi: 10.1186/s40814-022-01113-0. PMID 35897086
- [Derived] Grasaas E, Helseth S, Fegran L, Stinson J, Smastuen M, Haraldstad K. Health-related quality of life in adolescents with persistent pain and the mediating role of self-efficacy: a cross-sectional study. Health Qual Life Outcomes. 2020 Jan 30;18(1):19. doi: 10.1186/s12955-020-1273-z. PMID 32000787